CLINICAL TRIAL: NCT03812653
Title: Sleep for Stroke Management and Recovery Trial
Acronym: Sleep SMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); FusionHealth LLC (Unknown); Medical University of South Carolina (Other); University of Cincinnati (Other)
Responsible Party: Principal Investigator, Devin L. Brown, MD, Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00147316; 1U01NS099043-01A1 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Sleep Apnea; Sleep Apnea, Obstructive; Stroke; CPAP; Telemedicine; Home Sleep Apnea Test; Randomized Clinical Trial; Multicenter Trial
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Stroke

STUDY DESIGN:
Intervention Model Description: Intervention group receives automatically adjusting continuous positive airway pressure (CPAP) plus usual care.The control group receives usual care.
Who Masked: Outcomes Assessor
Masking Description: Eligible participants will be allocated in a 1:1 fashion to CPAP or no CPAP using a randomization method to protect subject treatment allocation and prevent potential selection biases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Arm: CPAP with Usual Care. (Experimental): 6 months of CPAP plus usual medical therapy.
  Interventions: Device: CPAP
- Control Arm: Usual Care. (No Intervention): 6 months of usual medical therapy alone.

INTERVENTIONS:
Device: CPAP — Automatically-adjusting continuous positive airway pressure (CPAP) delivered using a study supplied device.
  Arms: Intervention Arm: CPAP with Usual Care.

SUMMARY:
The purpose of this study is to determine whether treatment of obstructive sleep apnea (OSA) with positive airway pressure starting shortly after acute ischemic stroke (1) reduces recurrent stroke, acute coronary syndrome, and all-cause mortality 6 months after the event, and (2) improves stroke outcomes at 3 months in patients who experienced an ischemic stroke.

DETAILED DESCRIPTION:
Sleep SMART has a prospective, randomized, open-label, blinded-endpoint (PROBE) design. It is a multi-site, parallel-group superiority trial that compares 6 months of OSA treatment to usual care. The study includes two trials: a prevention study with an embedded recovery trial. 3062 subjects will be randomized over 5 years at 110 sites within the NINDS-funded StrokeNet clinical trials network.

ELIGIBILITY:
Current Inclusion Criteria, as of 6/28/2024:

1. Ischemic stroke within the prior 7 days.
2. NIH Stroke Scale Score ≥1 at the time of enrollment

Previous Inclusion Criteria, prior to 6/28/2024:

1. Ischemic stroke or TIA with ABCD ≥4, within prior 14 days.

Exclusion Criteria (for entire time period):

1. pre-event inability to perform all of own basic ADLs
2. unable to obtain informed consent from subject or legally authorized representative
3. incarcerated
4. known pregnancy
5. current mechanical ventilation (can enroll later if this resolves) or tracheostomy
6. current use of positive airway pressure, or use within one month prior to stroke
7. anatomical or dermatologic anomaly that makes use of CPAP interface unfeasible
8. severe bullous lung disease
9. history of prior spontaneous pneumothorax or current pneumothorax
10. hypotension requiring current treatment with pressors (can enroll later if this resolves)
11. other specific medical circumstances that conceivably, in the opinion of the site PI, could render the patient at risk of harm from use of CPAP
12. massive epistaxis or previous history of massive epistaxis
13. cranial surgery or head trauma within the past 6 months, with known or possible CSF leak or pneumocephalus
14. recent hemicraniectomy or suboccipital craniectomy (i.e. those whose bone has not yet been replaced), or any other recent bone removal procedure for relief of intracranial pressure
15. current receipt of oxygen supplementation >4 liters per minute
16. current contact, droplet, respiratory/airborne precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3062 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Time to Event Combined Outcome: new ischemic stroke, acute coronary syndrome, or all-cause mortality | 6 months post randomization
  The primary outcome is a time-to-event outcome defined as a participant having at least one of the following events within 6-months from randomization: new ischemic stroke, acute coronary syndrome or all-cause mortality
Modified Rankin Scale Score | 3 months post randomization
  Functional outcome as measured by the 9 question modified Rankin Scale (mRS-9Q). The mRS-9Q has 9 questions related to level of function. Outcomes range from 0 (no symptoms) to 6 (death).

SECONDARY OUTCOMES:
NIH Stroke Score (NIHSS) | 3 months post randomization
  Neurological outcome is measured by the NIHSS. The NIHSS scale ranges from 0 (no deficits) to 42.
Short Montreal Cognitive Assessment (MoCA) Score | 3 months post randomization
  Cognitive outcome is measured by the Short MoCA. The short MoCA is a 5 minute short version of the Montreal Cognitive Assessment (MoCA). This instrument tests phonemic verbal fluency (1 point), delayed recall (5 points), and orientation (6 points) with a score ranging from 0-12.
Quality of Life outcome | 3 months post randomization
  Quality of life outcome is measured by the shortened Stroke Specific Quality of Life Scale (SS-QOL). The short SS-QOL has 7 domains that include physical function, language, vision, thinking, energy, mood, and role function. There is 1 question from each domain. The 12 item SS-QOL is calculated by averaging the scores of these 12 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Devin Brown, MD, MS, Principal Investigator — University of Michigan; Ronald Chervin, MD, MS, Principal Investigator — University of Michigan
Locations (116):
- United States (116):
  - University of Alabama Hospital, Birmingham, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Dignity Health - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - TMC Healthcare, Tucson, Arizona
  - Banner- University Medical Center Tucson, Tucson, Arizona
  - Mercy San Juan Medical Center, Carmichael, California
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Scripps Memorial, La Jolla, California
  - UCSD Health La Jolla, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Doctors Medical Center of Modesto, Modesto, California
  - UCLA Kaiser Fontana, Ontario, California
  - UC Irvine, Orange, California
  - Casa Colina, Pomona, California
  - Kaiser Redwood, Redwood City, California
  - UC Davis Medical Center, Sacramento, California
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - Orange County Global Medical Center, Santa Ana, California
  - Olive View- UCLA Medical Center, Sylmar, California
  - John Muir Medical Center- Walnut Creek Campus, Walnut Creek, California
  - St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health, Fort Lauderdale, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - UF Jacksonville, Jacksonville, Florida
  - Brooks Rehabilitation Hospital, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Iowa Methodist, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton HealthCare, Louisville, Kentucky
  - Ochsner Medical Center - Main Campus, New Orleans, Louisiana
  - University Health Shreveport, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center,, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - Trinity Health Saint Mary's, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Mayo Clinic Saint Marys Campus, Rochester, Minnesota
  - Saint Cloud/Centracare Health, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Cox Medical Center, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - JFK Neuroscience Institute, Edison, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Hackensack Meridian Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Brooklyn, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Bellevue Hospital, New York, New York
  - NYU Langone -Tish Hospital Medical Center, New York, New York
  - NYP Columbia University Medical Center, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Suny Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center Atrium Health, Charlotte, North Carolina
  - Carolinas Rehab Northeast, Concord, North Carolina
  - Guilford Neurologic Associates, Inc, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - West Chester Hospital, West Chester, Ohio
  - St. John Health System, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - St. Luke's University Hospital Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - Penn State Milton S. Hershey Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Methodist University, Memphis, Tennessee
  - Baylor Scott & White Institute of Rehabilitation, Dallas, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Healthcare, Salt Lake City, Utah
  - The University of Vermont Medical Center Main Campus, Burlington, Vermont
  - UVA Medical Center, Charlottesville, Virginia
  - Inova Fairfax, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Ruby Memorial Hospital, Morgantown, West Virginia
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - University of Wisconsin University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
We will comply with the NIH Data Sharing Policy, Policy on the Dissemination of NIH-Funded Clinical Trial Information, the Clinical Trials Registration and Results Information Submission rule, and StrokeNet SOP on Network Data Sharing Policy. NDMC statisticians will generate data files from each data table and in compliance with HIPAA regulations each table will be de-identified. A minimum number of derived variables necessary to reproduce the primary analysis will be created. Within a year from acceptance of the primary manuscript or no later than two years from database lock, the public-use data sets will be submitted to the NINDS data repository along with final version of the study protocol, data dictionary and a user guide. Data along with signals from sleep apnea recordings will be submitted to the NHLBI National Sleep Research Resource.

REFERENCES:
- [Derived] Brown DL, Novitski K, Sickler JB, Hankla RM, Khattak F, Philpot E, Durkalski-Mauldin V, Sayyahmelli S, Patino C, Arevalo-Bermudez F, Roberts M, Sahelian A, Chervin RD. Use of a Generative Pretrained Transformer to Answer Questions and Facilitate a Large Randomized Controlled Trial. J Am Heart Assoc. 2025 Oct 21;14(20):e043333. doi: 10.1161/JAHA.125.043333. Epub 2025 Oct 21. PMID 41120814